CLINICAL TRIAL: NCT05401864
Title: Characteristics of Patients With Philadelphia Negative Myeloproliferative Neoplasms at Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ZeinabMekhemerTagBakr, Resident at Hematology Department , Principal Investigator, Assiut University
Other Study IDs: philadelphia negative MPNS
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Philadelphia Negative Myeloproliferative Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Classic Philadelphia chromosome-negative myeloproliferative neoplasms (MPNs) are a family of clonal chronic hematologic malignancies that include. polycythemia vera (PV), essential thrombocythemia (ET), and primary. Myelofibrosis (MF) . The classic MPNs historically have predominantly been diagnosed in older adults, with a median age at diagnosis of 60-72 years . Adults less than 40 years of age make up a largely underrepresented and therefore less studied subset of patients constituting 2.2-6.6% of yearly MPN cases in population- based study. These estimates are lower than incidence rate among patients between 40 and 49 years of age (9.1-10%), and have remained largely unchanged over the past four decades . However, with increasing trends in MPN incidence consequent to increased diagnostic recognition, better pathobiologic understanding, and more frequent JAK2/CALR/MPL mutational testing and newly revised WHO diagnostic criteria, it is conceivable that MPNs may be diagnosed at a higher frequency, in the younger patients, over time.

DETAILED DESCRIPTION:
Diagnosis of MPN according to the revised 2008 WHO criteria is based on a. combination of clinical, morphological, and molecular parameters ( Cardinal features of Philadelphia chromosome-negative MPN are increased red blood cell (RBC). production in PV, sustained thrombocytosis in ET, and bone marrow (BM) fibrosis in PMF. Molecular markers, such as JAK2 V617F, JAK2 exon 12, and MPL mutations, have increased our knowledge of the pathogenesis of MPNs as well as the accuracy of diagnosis. Furthermore, many recent studies have reported that the calreticulin mutation (mutation in exon 9 of CALR) is found in the majority of patients with MPN with non mutated JAK2 . There are many controversies with regard to the subjectivity and the lack of reproducibility of the histological criteria. And BM assessment is not always needed, especially in PV. However, histologic evaluation of the pathologic features of megakaryocytic, granulocytic, and erythroid series and cellularity is important in differentiating MPNs, especially ET and PMF . Sometimes, patients with occult MPN present with normal blood counts because of gastrointestinal bleeding and associated iron deficiency, splenomegaly, or simply because they are in an early stage of the disorder . In cases of clinically suspicious MPN, such as intra-abdominal thrombosis with normal blood counts, careful investigation is needed.

diagnostic criteria for myeloproliferative (World Health Organization) 2008. Polycythemia refers to an increase in the number of red blood cells in the body. The extra cell cause the blood to be thicker, and this, in turn, increases the risk of other health issues, such as blood clots.

Maior criteria including. Hemoglobin > 18.5 g/dL (men), > 16.5 g/dL (women) or Presence of JAK2 V617F or JAK2 exon 12 mutation Minor criteria: BM hypercellularity with trilineage myeloproliferation Subnormal serum erythropoitin. Endogenous erythroid colony formation in vitro.

Management of polycythemia: The most common treatment for polychythemia vera is having frequent blood withdrawals, using a needle in a vein (phlebotomy).

Drugs that reduce the number of red blood cells If phlebotomy alone doesn't help enough, your doctor may suggest medications that can reduce the number of red blood cells in your bloodstream. Examples include: Hydroxyruea (Droxia, Hydrea), Interferon alfa-2b (Intron A), Ruxolitinib (Jakafi), Busulfan (Busulfex, Myleran) .

Primary myelofibrosis (PMF) is a rare bone marrow disorder that is characterized by abnormalities in blood cell production (hematopoiesis) and scarring (formation of fibrous tissue) within the bone marrow. Bone marrow is the soft, spongy tissue that fills the center of most bones. Major criteria including. Megakaryocyte proliferation and atypiab, accompanied by either reticulin and/or collagen fibrosis, orc Not meeting WHO criteria for PV, CML, MDS, or other myeloid neoplasm Demonstration of JAK2 V617F or other clonal marker or no evidence of bone marrow fibrosis.

prognosis scoring was the international prognostic scoring system (IPSS). IPSS was first produced in 2009 and was designed for application at the time of diagnosis. This IPSS was the result of data from 1054 consecutively diagnosed patients with PMF from 1980 to 2007. 4 risk groups were identified, with median survivals ranging from 23 years (high-risk) to 11.3 months (low-risk). Abnormal cytogenetic findings did not appear to affect patient outcomes. IPSS included five risk factors: age >65 years, hemoglobin <10 g/dl, leukocyte count >25 x 109/L, circulating blasts ≥1% and constitutional symptoms. In 2010, DIPSS was adapted from IPSS, which allowed clinicians to use prognostic scoring at any time in the clinical course. Both IPSS and DIPSS (Dynamic IPSS) used the same five clinical risk factors to determine patient prognosis.

Management of mylofibrosis: Low-risk myelofibrosis may not require immediate treatment, while people with high-risk myelofibrosis may consider an aggressive treatment, such as bone marrow transplant. For intermediate-risk myelofibrosis, treatment is usually directed at managing symptoms. Immediate treatment may not be necessary Myelofibrosis treatment may not be necessary if you aren't experiencing symptoms. You might not need treatment right away if you don't have an enlarged spleen and you don't have anemia or your anemia is very mild. Rather than treatment, your doctor is likely to monitor your health closely through regular checkups Treatments for anemia: Blood transfusions, Androgen therapy, Thalidomide and related medications.

Treatments for an enlarged spleen: Chemotherapy, Targeted drug therapy, (splenectomy). If your spleen becomes so large, Radiation therapy. Bone marrow transplant.

Essential thrombocytosis (ET), or primary thrombocythemia, is a rare disorder in which the body produces too many platelets for unknown reasons. This can cause abnormal blood clotting or bleeding. Majorcriteria: Sustained platelet count > 450 × 109/LProliferation of megakaryocytes with enlarged, mature morphology Not meeting WHO criteria for PV, PMF, CML, MDS or other myeloid neoplasm Demonstration of JAK2 V617F or other clonal marker, or no evidence for reactive Thrombocytosis. Patients with low-risk ET are usually managed with low-dose aspirin, whereas treatment of high-risk ET is based on the use of cytoreductive therapy, with hydroxyurea as the drug of choice and IFN-α being reserved for young patients or pregnant women

ELIGIBILITY:
Inclusion Criteria:

- Patients with Philadelphia negative above 18yrs old who were attend at our unit over 2 years duration.

Exclusion Criteria:

* All pt with Philadelphia positive and below 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Philadelphia negative myloproliferative neoplasms at Assuit university hospital
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
characteristics data of philadilphia negative myloproleferative neoplasm | 2 years
  Characteristics data of philadilphia negative myloproleferative neoplasm admitted inassiut university hospital in 2years in single center experience this data including age .sex ipss score and management of MPN

REFERENCES:
- [Background] Tefferi A, Pardanani A. Myeloproliferative Neoplasms: A Contemporary Review. JAMA Oncol. 2015 Apr;1(1):97-105. doi: 10.1001/jamaoncol.2015.89. PMID 26182311
- [Background] Tefferi A. Primary myelofibrosis: 2017 update on diagnosis, risk-stratification, and management. Am J Hematol. 2016 Dec;91(12):1262-1271. doi: 10.1002/ajh.24592. PMID 27870387
- [Background] Srour SA, Devesa SS, Morton LM, Check DP, Curtis RE, Linet MS, Dores GM. Incidence and patient survival of myeloproliferative neoplasms and myelodysplastic/myeloproliferative neoplasms in the United States, 2001-12. Br J Haematol. 2016 Aug;174(3):382-96. doi: 10.1111/bjh.14061. Epub 2016 Apr 7. PMID 27061824
- [Background] Barbui T, Thiele J, Carobbio A, Passamonti F, Rumi E, Randi ML, Bertozzi I, Vannucchi AM, Gisslinger H, Gisslinger B, Finazzi G, Ruggeri M, Rodeghiero F, Rambaldi A, Gangat N, Tefferi A. Disease characteristics and clinical outcome in young adults with essential thrombocythemia versus early/prefibrotic primary myelofibrosis. Blood. 2012 Jul 19;120(3):569-71. doi: 10.1182/blood-2012-01-407981. Epub 2012 Jun 13. PMID 22700720
- [Background] Szuber N, Vallapureddy RR, Penna D, Lasho TL, Finke C, Hanson CA, Ketterling RP, Pardanani A, Gangat N, Tefferi A. Myeloproliferative neoplasms in the young: Mayo Clinic experience with 361 patients age 40 years or younger. Am J Hematol. 2018 Dec;93(12):1474-1484. doi: 10.1002/ajh.25270. Epub 2018 Sep 27. PMID 30157297
- [Background] Andrikovics H, Krahling T, Balassa K, Halm G, Bors A, Koszarska M, Batai A, Dolgos J, Csomor J, Egyed M, Sipos A, Remenyi P, Tordai A, Masszi T. Distinct clinical characteristics of myeloproliferative neoplasms with calreticulin mutations. Haematologica. 2014 Jul;99(7):1184-90. doi: 10.3324/haematol.2014.107482. Epub 2014 Jun 3. PMID 24895336
- [Background] Barbui T, Barosi G, Birgegard G, Cervantes F, Finazzi G, Griesshammer M, Harrison C, Hasselbalch HC, Hehlmann R, Hoffman R, Kiladjian JJ, Kroger N, Mesa R, McMullin MF, Pardanani A, Passamonti F, Vannucchi AM, Reiter A, Silver RT, Verstovsek S, Tefferi A; European LeukemiaNet. Philadelphia-negative classical myeloproliferative neoplasms: critical concepts and management recommendations from European LeukemiaNet. J Clin Oncol. 2011 Feb 20;29(6):761-70. doi: 10.1200/JCO.2010.31.8436. Epub 2011 Jan 4. PMID 21205761
- [Background] Tefferi A, Vardiman JW. Classification and diagnosis of myeloproliferative neoplasms: the 2008 World Health Organization criteria and point-of-care diagnostic algorithms. Leukemia. 2008 Jan;22(1):14-22. doi: 10.1038/sj.leu.2404955. Epub 2007 Sep 20. PMID 17882280
- [Background] Klampfl T, Gisslinger H, Harutyunyan AS, Nivarthi H, Rumi E, Milosevic JD, Them NC, Berg T, Gisslinger B, Pietra D, Chen D, Vladimer GI, Bagienski K, Milanesi C, Casetti IC, Sant'Antonio E, Ferretti V, Elena C, Schischlik F, Cleary C, Six M, Schalling M, Schonegger A, Bock C, Malcovati L, Pascutto C, Superti-Furga G, Cazzola M, Kralovics R. Somatic mutations of calreticulin in myeloproliferative neoplasms. N Engl J Med. 2013 Dec 19;369(25):2379-90. doi: 10.1056/NEJMoa1311347. Epub 2013 Dec 10. PMID 24325356
- [Background] Nangalia J, Massie CE, Baxter EJ, Nice FL, Gundem G, Wedge DC, Avezov E, Li J, Kollmann K, Kent DG, Aziz A, Godfrey AL, Hinton J, Martincorena I, Van Loo P, Jones AV, Guglielmelli P, Tarpey P, Harding HP, Fitzpatrick JD, Goudie CT, Ortmann CA, Loughran SJ, Raine K, Jones DR, Butler AP, Teague JW, O'Meara S, McLaren S, Bianchi M, Silber Y, Dimitropoulou D, Bloxham D, Mudie L, Maddison M, Robinson B, Keohane C, Maclean C, Hill K, Orchard K, Tauro S, Du MQ, Greaves M, Bowen D, Huntly BJP, Harrison CN, Cross NCP, Ron D, Vannucchi AM, Papaemmanuil E, Campbell PJ, Green AR. Somatic CALR mutations in myeloproliferative neoplasms with nonmutated JAK2. N Engl J Med. 2013 Dec 19;369(25):2391-2405. doi: 10.1056/NEJMoa1312542. Epub 2013 Dec 10. PMID 24325359